CLINICAL TRIAL: NCT03270592
Title: Assessment of Service and Hearing Dogs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Collaborators: Ministry of Health and Social Affairs, Sweden (Other Government)
Responsible Party: Principal Investigator, Martina Lundqvist, Principal Investigator, Linkoeping University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Dnr 157-09
Record Dates: First submitted 2017-08-31; First posted 2017-09-01 (Actual); Last update posted 2017-09-05 (Actual); Status verified 2017-09

CONDITIONS: Impairment; Diabetes; Epilepsy
Keywords: Service dogs; Alert dogs; Costs; Quality of Life; Cost-effectiveness
MeSH Terms: conditions — Diabetes Mellitus; Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Service dogs (Other): Single arm study using a before after design where Before represent having a regular companion dog and after represent having a certified service dog
  Interventions: Other: Service dog

INTERVENTIONS:
Other: Service dog — Use of a individualized certified service dog

SUMMARY:
For persons with impairments and certain illnesses the use of service dogs may have positive effect. The effects of using these dogs to assist in every day life need to be studied further.The aim of the study was to assess how health care consumption was effected by using certified service dogs and to study the cost-effectiveness of having a certified service dog.

DETAILED DESCRIPTION:
This is an exploratory before and after study with the aim to study how health care consumption was effected by using certified service dogs and to study the cost-effectiveness of having a certified service dog. Data was collected before the education of the dog started and the follow-up was made three months after completion of the education. Data was collected on Health care consumption and outcomes in terms Health related quality of life and Health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age over 16 years
* Having a regular companion dog
* Being in need of a certified service dog (due to impairment, diabetes, epilepsy and deafness)

Exclusion Criteria:

* Psychiatric illness

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2009-09-17 (Actual); Primary Completion 2014-07-02 (Actual); Study Completion 2014-07-02 (Actual)

PRIMARY OUTCOMES:
Total costs | Three months follow-up
  Health care costs, cost of informal care, municipal costs
Health related quality of life, EQ-5D | Tree months follow-up
  EQ-5D is a generic quality of life instrument including five dimensions

SECONDARY OUTCOMES:
Cost-effectiveness | Life time perspective
  Cost per quality adjusted life years (QALY)
Health related quality of life, RAND-36 | Three months follow-up
  RAND-36 is a generic quality of life instrument including eight dimensions
WHO-5 wellbeing index | Three months follow-up
  WHO-5 wellbeing index is an index measuring wellbeing on five dimensions
Rosenberg self-esteem scale | Three month follow-up
  Rosenberg self-esteem scale measures self esteem with ten questions
EQ-VAS | Three months follow-up
  EQ-VAS is a Visual analogue scale ranging from 0 to 100 (perfect Health)

CONTACTS AND LOCATIONS:
Overall Officials: Lars-Åke Levin, Professor, Study Director — Linkoeping University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lundqvist M, Levin LA, Roback K, Alwin J. The impact of service and hearing dogs on health-related quality of life and activity level: a Swedish longitudinal intervention study. BMC Health Serv Res. 2018 Jun 27;18(1):497. doi: 10.1186/s12913-018-3014-0. PMID 29945630